CLINICAL TRIAL: NCT02377934
Title: Evaluation of Radiation Induced Pulmonary Hypertension Using MRI in Stage III NSCLC Patients Treated With Chemoradiotherapy. A Pilot Study
Acronym: MRI-HART
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RT2011-02
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Cardiac MRT; Radiotherapy
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Cardiac Magnetic Resonance Imaging (MRI)

SUMMARY:
In the radiotherapeutic treatment of lung cancer, the dose that can be safely applied to the tumour is limited by the risk of radiation induced lung damage. This damage is characterized by parenchymal damage and vascular damage. In rats, we have found that radiation-induced vascular damage results in increased pulmonary artery pressure. Interestingly, the consequent loss of pulmonary function could be fully explained by this increase in pulmonary artery pressure. We hypothesize that also in patients a radiation induced increase in pulmonary artery pressure can be observed after radiotherapy, which may contribute to the development of radiation pneumonitis.

The objective is to test the hypothesis that radiotherapy for lung cancer induces an increase in pulmonary artery pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* WHO PS 0-2
* Histological or cytological confirmation of non-small cell lung cancer or an 18F-FDG-positive, growing mass on CT-thorax suggestive of NSCLC.
* Stage IIIA or IIIB
* Patients with extensive mediastinal lymph node involvement (such as N3), or large primary tumour size
* Adequate pulmonary function estimated by flow volume curves
* Life expectancy of at least 6 months
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol; those conditions should be discussed with the patient before registration in the trial.
* Planned for 25 x 2.4 Gy, with concomitant chemotherapy
* Before patient registration, written informed consent will be obtained.

Exclusion Criteria:

* Presence of contra-indications for undergoing MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with stage III NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in pulmonary artery pressure | 6 and 12 weeks after completion chemoradiotherapy

SECONDARY OUTCOMES:
Pulmonary artery velocity; right ventricle (RV) dimensions and RV-function | 6 and 12 weeks after completion chemoradiotherapy
The assessment of RV-dimensions and RV-function | 6 and 12 weeks after completion chemoradiotherapy
The incidence of clinical signs of radiation pneumonitis according to SWOG-criteria | 6 weeks after completion treatment
The incidence of radiological signs of pulmonary fibrosis according to CTCAE4.0 | 12 weeks after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robin Wijsman, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands